CLINICAL TRIAL: NCT02512627
Title: Evolving Methods to Combine Cognitive and Physical Training for Individuals With Mild Cognitive Impairment: An Efficacy Study
Brief Title: Evolving Methods to Combine Cognitive and Physical Training for Individuals With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103-6651A3
Record Dates: First submitted 2015-07-20; First posted 2015-07-31 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-05

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; exercise; cognitive training
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Cognitive Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive training group (Cog) (Active Comparator): The BrainHQ program will be used to train different cognitive functions of the participants. The participants will practice tasks that involve the abilities of visuospatial processing, attention, memory, language, and/or executive functions. The tasks will become more difficult as the participants progress in their abilities.
  Interventions: Behavioral: Cognitive training
- Physical exercise group (PE) (Active Comparator): The participants in this group participate in multimodal exercise programs including aerobic exercise, balance, and strength training. The entire exercise program for the PE group will contain 10 minutes of warm-up, 70 minutes of physical exercise, and 10 minutes of cool-down. The 70 minutes of exercise session will be break up into 2 to 3 parts, and the participants can rest as needed during the exercise period.
  Interventions: Behavioral: Physical exercise
- Sequential training group (Seq) (Experimental): The participants in this group will first perform 45 minutes of physical exercise followed by 45 minutes of cognitive training. The physical exercise training will be similar to the programs used in the PE group. The entire exercise program for the PE group will contain 5 minutes of warm-up, 35 minutes of physical exercise, and 5 minutes of cool-down. The cognitive training will be implemented with BrainHQ similar to what has been described in the COG group.
  Interventions: Behavioral: Cognitive training; Behavioral: Physical exercise
- Dual-task training group (Dual) (Experimental): In this group, the participants will be instructed to perform physical exercise and cognitive tasks simultaneously (e.g., math calculation while stepping). The difficulty of the cognitive tasks will increase as the participants improve in their performance.
  Interventions: Behavioral: Cognitive training; Behavioral: Physical exercise

INTERVENTIONS:
Behavioral: Cognitive training — visuospatial, attention, memory, and executive abilities
  Arms: Cognitive training group (Cog); Dual-task training group (Dual); Sequential training group (Seq)
Behavioral: Physical exercise — endurance, balance, and mobility
  Arms: Dual-task training group (Dual); Physical exercise group (PE); Sequential training group (Seq)

SUMMARY:
This study aims to investigate and compare the intervention effects of combining exercise and cognitive training (either sequentially or simultaneously in a dual-task paradigm) in elderly with mild cognitive impairment. The investigators hypothesize that (1) both sequential and dual-task training can induce greater improvements in the outcome measures than single mode of training; (2) the improvement in cognitive functions and other outcomes may differ between the groups.

DETAILED DESCRIPTION:
Background and study aims:

Mild cognitive impairment (MCI) or minor neurocognitive disorder is a syndrome defined as an intermediate stage between cognitively intact and clinically diagnosed dementia. The age-adjusted prevalence of MCI in Taiwan is approximately 18%, while women have higher prevalence for MCI than men. The progression rate from MCI to dementia ranges from 10 to 15% each year, and over 50% of the MCI population will develop into severe cognitive impairment or dementia in 5 years. Therefore, early detection of the individuals who manifest MCI and provide appropriate interventions may help reduce the burden of their caregivers and the medical expenses of the health-care system. Previous studies found that cognitive training or exercise has emerged as an important therapeutic approach for individuals with MCI. However, the intervention effects of combining exercise and cognitive training remain to be determined. Furthermore, whether exercise and cognitive training should be administered in sequential order or simultaneously is an important question to pursue. The overall goal of this study is to determine and compare the intervention effects cognitive training, exercise, and combining cognitive and exercise training in individuals with MCI.

Who can participate? Individuals with MCI.

What does the study involve? The participants will receive a total of 36 training sessions, and each session will contain 90 minutes of training. Training frequency will be 2-3 times per week for 12-18 weeks. All participants will received pretreatment test, post treatment test, and a 6-month follow-up test.

What are the possible benefits and risks of participating? The possible benefits include improvement in cognitive, physical, and daily functions. There are no risks for participating.

Where to conduct the study? The investigators anticipate recruiting a total of 80 participants from geriatric day care centers and nursing homes from multiple cities in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. able to follow instruction,
2. clinical dementia rating (CDR) = 0.5 or 1,
3. self- or informant-reported memory or cognitive complaint, and
4. able to perform activities of daily living (Barthel Index ≥ 70).

Exclusion Criteria:

1. recent myocardial infarction,
2. heart failure,
3. recent heart surgery,
4. severe asthma,
5. concomitant with other neurological disorders, or
6. joint deformity that might prevents them performing exercise or cognitive training.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Change scores of Montreal Cognitive Assessment (MoCA) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The MoCA will be used to assess general cognitive functions. It examines several cognitive domains with a total score of 30.
Change scores of Stroop test | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Stroop test will be used to assess the processing speed, inhibition, set-shifting, and selective attention abilities. The participants will be tested under 2 conditions: congruent and incongruent conditions. In the congruent condition, the color ink of a word is consistent with the written color name; while the color ink differs from the written color name under the incongruent condition.
Change scores of Dual-task test | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The dual-task tests will be assessed to determine the ability for an individual to perform 2 tasks simultaneously. The investigators will assess the dual-task performance during walking and performing box and block test. The results of the dual-task tests will provide information regarding to whether the 2 tasks compete for the same class of neural resources or one of the tasks can be carried out automatically.
Change scores of Timed up and go (TUG) test | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The TUG test will be used to assess the mobility and dynamic balance ability. The participants will be required to stand up from a chair, walk 3 meters, turn around, then walk back to the chair, and sit down. The time to complete the TUG test has been shown to be a good indicator to detect potential fallers and frail elderly (Podsiadlo & Richardson, 1991). The test-retest reliability of TUG on individuals with cognitive impairment was excellent (Blankevoort, van Heuvelen, & Scherder, 2013).

SECONDARY OUTCOMES:
Change scores of the Verbal Fluency Test | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  Verbal fluency tests will be used to evaluate the semantic memory of the participants. The participants will be instructed to say as many words as possible from a given category (i.e., fruit or animal) in 1 minute. The validity, reliability, and normative performance of verbal fluency tests have been well-established (Harrison, Buxton, Husain, & Wise, 2000).
Change scores of the Useful Field of View (UFOV) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  Useful field of view (UFOV) is the visual area over which useful information could be obtained at a quick glance without eye or head movements. This UFOV will be assessed with the BrainHQ program. The UFOV will assess the abilities of visuomotor processing speed, divided attention, and selective attention (Ball, Edwards, & Ross, 2007).
Change scores of the 30 second chair stand test (CST) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The 30 second chair stand test (CST) will be assessed to indicate the strength and endurance level of the lower extremities. The participants will be asked to stand up from a standardized chair and then sit down as many times as possible within 30 seconds. The feasibility and reliability of using CST in people with cognitive impairment have been established to be good (Blankevoort et al., 2013).
Change scores of the Chinese version of the International Physical Activity Questionnaires (IPAQ) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Chinese version of the International Physical Activity Questionnaires (IPAQ) is an international measure for health-related physical activity. A short form of IPAQ will be used to assess changes in physical activity before and after intervention in this study. The reliability and validity of IPAQ has been established across 12 countries (Craig et al., 2003).
Change scores of the Barthel Index (BI) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  Assess activities of daily living
Change scores of the Lawton Instrumental Activities of Daily Living Scale | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  Assess activities of daily living.
Change scores of the Disability Assessment for Dementia (DAD) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  Assess activities of daily living.
Change scores of the Quality of Life in Alzheimer's Disease Instrument (QoLAD) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Chinese version of QoLAD will be used.
Change scores of the Caregiver Burden Inventory (CBI) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Chinese version of CBI will be used.
Change scores of the Geriatric Depression Scale (GDS) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The Chinese version of short form GDS will be used.
Change scores of the Community Integration Questionnaire (CIQ) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The CIQ measures items relevant to home integration, social integration, and productive activities.
Change scores of the ActiGraph GX3 accelerometers Change scores of the ActiGraph | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The actigraphy will be placed on the waist for a 3-day period immediately before and after the intervention. The participants will wear the actigraphy during all daily activities except for those that involve water (i.e., showering or swimming).
Change scores of evaluating isometric knee flexors and extensors muscle strength | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The participant will be seated upright in a chair with back support, the knee will be placed in 90-degree flexion and the evaluator will stabilize the thing to eliminate synergistic movements. Participants will be asked to perform a maximal isometric contraction of knee flexion and extension with both lower extremities. The investigators will record the mean value of 3 attempts.
Change scores of using hand dynamometer to measure grip strength of both hand | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The participant is seated, with the elbow at 90-degree flexion. The investigators will record the mean value of 3 attempts.
Change scores of Wechsler Memory Scale - Third Edition (WMS-III) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The investigators will use the WMS-III subtests, including Faces Recognition (score range 0-48), Verbal Paired Associates (score range 0-32), Word Lists (0-48), and Spatial Span (0-32) to assess the immediate, delayed, and working memory tests. Higher scores indicated better performance for each subtest. The raw score of each subtest will also be transferred to standardized Z scores and summed to represent an index of general memory function.
Change scores of Wechsler Adult Intelligence Scale - Third Edition (WAIS-III) | baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The WAIS-III includes tests that evaluate cognitive functions in verbal comprehension, working memory, perceptual organization, and processing speed. The subtests that the investigators will use are the Digit Symbol-Coding (scores range 0-133) and Matrix Reasoning tests (0-26). The raw score of each subtest will also be transferred to standardized Z scores and summed to represent an index of general cognitive function.
BDNF val66met genotype | baseline
  Saliva samples will be collected at baseline to determine the Brain-Derived Neurotrophic Factor (BDNF) val66met genotype.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yi Wu, ScD, Principal Investigator — Chang Gung Memorial Hospital
Locations (9):
- Taiwan (9):
  - Baliexcelsior Nursing Home, New Taipei City
  - Pine nursing home, Taichung
  - Zhishan community home, Taipei
  - Bailing clinics and nursing homes, Taipei
  - Shihlin cum day care center, Taipei
  - Xihu day care center, Taipei
  - TaoSheng Nursing home, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
  - Chang Gung Memorial Hospital Taoyuan Branch, Taoyuan District

REFERENCES:
- [Derived] Lee YY, Wu CY, Teng CH, Hsu WC, Chang KC, Chen P. Evolving methods to combine cognitive and physical training for individuals with mild cognitive impairment: study protocol for a randomized controlled study. Trials. 2016 Oct 28;17(1):526. doi: 10.1186/s13063-016-1650-4. PMID 27793183